CLINICAL TRIAL: NCT06657339
Title: National Registry of Obesity Treatment by Endosleeve
Status: Not yet recruiting | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, VANBIERVLIET, Director, Head of Endocopy, Principal Investigator, Medical doctor, Société Française d'Endoscopie Digestive
Other Study IDs: SFED-153
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: Endosleeve; Endoscopic gastroplasty; Endoscopic suture
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic sleeve gastroplasty: Therapeutic endoscopy using a gastric suturing device (OverStitch™/Endomina™) according to the practices of the investigating center
  Interventions: Procedure: Therapeutic endoscopy endosleeve using a gastric suturing device (OverStitch™/Endomina™)

INTERVENTIONS:
Procedure: Therapeutic endoscopy endosleeve using a gastric suturing device (OverStitch™/Endomina™) — The patient will undergo therapeutic endoscopy under general anesthesia, either as outpatient or inpatient care, based on the recommendations of the investigating physician, taking into account anesthetic risks and comorbidities. Two CE-marked gastric suturing devices may be used at the discretion of the investigating center based on their practices
  OverStich™ allows for tissue fixation via a gastroscope, creating a durable suture through a transabdominal fixation technique. The procedure lasts about 45 minutes and includes measures to prevent vomiting.
  Endomina™ is a single-use device that captures the gastric mucosa to create successive plications, allowing for effective suturing along the greater curvature of the stomach.

SUMMARY:
Obesity and overweight have emerged as public health problems of a pandemic nature, significantly reducing the life expectancy of those affected. Obesity has a considerable medico-economic impact, linked to the treatments it requires and its comorbidities. Currently, the prevention of obesity in our Western societies is not effective enough, as the prevalence and incidence of obesity and overweight continue to rise worldwide. In France, the therapeutic management of this condition is governed by the HAS and is summarized as a surgical approach for type 2 obesity with comorbidity or type 3 obesity, with three authorized methods that have shown sufficient evidence: gastric banding, sleeve gastrectomy (or longitudinal sleeve gastrectomy), and Roux-en-Y gastric bypass.

With the advent of organ-preserving interventional endoscopy, the systematic use of these surgical methods, although effective for total weight loss and excess weight loss, raises questions. Indeed, these new therapeutic endoscopic approaches, which are less invasive, less costly, and respectful of anatomy, currently show convincing cohort results in the short term (12 to 24 months) and require confirmation of their effectiveness and safety in the long term (5 years) so that they can become first-line therapeutic methods in the near future. At the request of the HAS in its self-referral of 2020 and then in 2022, this prospective registry aims to confirm the effectiveness and safety of the endosleeve (or endoscopic sleeve) in the long-term therapeutic management of obesity within the framework of everyday practice in national reference centers for obesity treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Patient with a body mass index (BMI) ≥ 30 kg/m²;
* Signed informed consent

Exclusion Criteria:

* Contraindication to performing an upper endoscopy or using an endoscopic plication system according to the instructions for use (IFU);
* Presence of an ulcer in the gastric body or fundus;
* Achalasia, severe esophagitis (Los Angeles grade C or D);
* ENT or esophageal malformation;
* Gastrointestinal disease (including stenosis), history of previous gastric surgery (including bariatric surgery, previous endoscopic gastroplasty);
* Congestive gastropathy, gastric polyposis, gastric or esophageal varices, risk of gastric tumor disease due to personal or family history;
* Positive Helicobacter pylori status with failed eradication treatments;
* Uncontrolled or severe eating disorder or psychiatric illness;
* Substance abuse or chronic alcoholism;
* Severe renal insufficiency (stage 4 or 5), Cirrhosis Child B or C;
* Anticoagulant or antiplatelet treatment that cannot be stopped or replaced according to international recommendations (ESGE 2021);
* Coagulation or hemostasis disorders (PT < 60%, platelets < 60,000/mm³);
* Mental deficiency of the subject making participation in the trial impossible;
* Patient not affiliated with a social security scheme;
* Pregnant women, breastfeeding individuals;
* Inability to understand or sign the informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any referred patient with obesity and a BMI > 30 kg/m² who meets the inclusion criteria and is considered suitable for therapeutic management of obesity will be invited to participate in the study at the investigating centers
Sampling Method: Non-Probability Sample
Enrollment: 354 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of total weight loss (TWL) in % 5 years afther endosleeve | 5 years
  To determine the proportion of patients who met the PIVI criteria after endosleeve without additional techniques

SECONDARY OUTCOMES:
Measurement of total weight loss (TWL) in % | 12 et 24 months
  Determine total weight loss (TWL) afther endosleeve at 12, 24 months,
Measurement excess weight loss after the endosleeve intervention. | 12, 24 months, and 5 years
  Determine excess weight loss (EWL) after the endosleeve intervention, with positivity established by the PIVI criteria (EWL > 25% at 12 months), and evaluate the long-term evolution of this EWL
Measurement of the percentage of postoperative complications according to the AGREE classification | Day 1 and Day 30.
  The safety of this procedure will be evaluated by recording complications perioperatively (Day 1) and post-procedure (Day 30) according to the AGREE criteria and using the PIVI criteria (positive if the complication rate is < 5%).
Measurement of remission (or regression) of pre-existing comorbidities | 12 months, 24 months, and 5 years.
  Determine the impact on pre-existing metabolic comorbidities :
  1. Diabetes remission = HbA1C < 6.5%, 3 months after discontinuation of all treatment / Regression or improvement of diabetes involving a decrease of more than 0.5% in HbA1C according to recognized criteria
  2. Hypertension = Systolic blood pressure (SBP) < 140 mmHg and/or Diastolic blood pressure (DBP) < 90 mmHg without any treatment / Decrease in the number of therapeutic classes;
  3. Obstructive Sleep Apnea Syndrome (OSAS) = Number of apneas less than 5 without equipment / Decrease in OSAS stage = mild (5 to 15 per hour), moderate (15 to 30), or severe (more than 30) with or without equipment;
  4. Steatohepatitis = quantification by MRI of the % of fat in the liver with a decrease of more than 30%;
  5. Dyslipidemia = normalization or improvement of LDL cholesterol and triglyceride levels without the addition of new drug therapies.
Occurrence of metabolic comorbidities | 12 months, 24 months, and 5 years
  The occurrence of metabolic comorbidities such as diabetes, hypertension (HTN), obstructive sleep apnea syndrome (OSAS), steatohepatitis, and dyslipidemia will be assessed at 12, 24 months, and at the end of the follow-up period. Each comorbidity will be evaluated according to its specific definitional criteria
Outpatient procedures | 30 days
  Number of outpatient procedures performed without the need for readmission within 30 days of follow-up
Bariatric procedures performed following the initial intervention | Day 1 and Day 30.
  Number and type of bariatric procedures performed following the initial intervention (Redo EndoSleeve, medication treatment such as GLP-1 agonists or equivalent, instrumental treatment with a balloon or other methods)
Conversion rates in bariatric surgery and their feasibility | 3 years and 5 years
  Number of conversions to bariatric surgery (Sleeve and bypass) and their feasibility (whether the procedure was possible)
Predictive factors for response, weight regain, and plateau at the EndoSleeve | 3 months, 6 months and 1 year
  Determination of predictive factors for response, failure (<5% total weight loss at 6 months), weight regain (50% of the lost weight regained at or after one year), and plateau with EndoSleeve (≥10% weight loss but no further loss for more than 3 months)
Sequence of bariatric procedures that led to the best weight response | 5 years
  Description of the sequence of bariatric procedures leading to the best weight loss outcome after 5 years of follow-up
Measurement of the improvement in quality of life. | 12 months , 24 months, and at 5 years of follow-up.
  Impact on quality of life will be measured through quality of life questionnaires (BAROS questionnaire) before the intervention and during each medical visit, to assess psychological health before and after the intervention.